CLINICAL TRIAL: NCT01478672
Title: Medium Term Health Coaching and Life-long Monitoring in Cardiovascular Disease in Norrbotten
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luleå Tekniska Universitet (Other)
Collaborators: County Council of Norrbotten, Sweden (Other Government)
Responsible Party: Principal Investigator, Inger Lindberg, Investigator, Luleå Tekniska Universitet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LTU-Medium health coaching
Record Dates: First submitted 2011-11-02; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes; Heart Disease; Quality of Life
Keywords: Promotion health
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention)
- Health coaching and and Life-long Monitoring (Experimental)
  Interventions: Procedure: Health Coaching and Life-long Monitoring

INTERVENTIONS:
Procedure: Health Coaching and Life-long Monitoring — Participants receive tablet PCs with software that collects and transmit diagnostic measurements. Measurements are performed by the participants following indications of the health coaching team. Equipment used by all participants: • blood pressure meter, • pedometer • pulse watch• 2-channel electrocardiograph. Measured values are entered manually by the participants, unrealistic values are refused and values are provided with a time-stamp. Measurements is reviewed in a graphical display. Measured values are accessed by the health coaching team that develops an individualized measurement and medication scheme. Reminders are provided by the software and can be exported to personal calendars or mobile phones. Secure authentication of users is be provided
  Arms: Health coaching and and Life-long Monitoring

SUMMARY:
The purpose of this study is to evaluate whether the introduction of large-scale personalized and technology supported telemonitoring and health coaching interventions produces benefits in terms of health related quality of life, health status and empowerment of patients with a cardiovascular disease. In addition, the trials evaluate the economical and organizational impact of the new services and examine their acceptability by patients and health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of arterial hypertension ischemic heart disease,
* atrial fibrillation or other arrhythmia,
* congestive heart failure (study heart disease)
* HbA1C > 53mmol/mol (study diabetes)
* Age > 18 years
* Capability of filling in questionnaires in the own language
* Capability to use the devices provided
* Being cognitively able to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
SF-36 | 12 months follow-up
  Questionnaire, 36 questions ref Ware, 2000 version 2

SECONDARY OUTCOMES:
HbA1c (for patients with type-2D) Blood pressure for patient with heart disease | 12 months follow-up
  HbA1c is a long-term sugar / serum glucose test, it is a blood test that gives a measure of blood sugar levels two to three months before sampling.
Bloodpressure | 12 months follow-up
Blood lipids | 12 months follow-up
Bodyweight | 12 months follow-up
Smoking habits | 12 months follow-up
Alcohol consumption | 12 months follow-up
SOC-13 | 12 months follow-up
  SOC-13 (sense of coherence, SOC) is a term that reflects the ability to cope with stress and is the essence of the salutogenic theory of health. SOC consists of three subordinate concepts, manageability, meaningfulness and comprehensibility.
EQ-5D | 12 monts follow-up
  EQ5D (5d) is a standardized instrument to measure and describe health outcomes. It can be used to measure health at the individual level in clinical settings and to measure a population's health locally and nationally.

CONTACTS AND LOCATIONS:
Locations (1):
- Luleå University of Technology, Luleå, Sweden

REFERENCES:
- [Derived] Lindberg I, Torbjornsen A, Soderberg S, Ribu L. Telemonitoring and Health Counseling for Self-Management Support of Patients With Type 2 Diabetes: A Randomized Controlled Trial. JMIR Diabetes. 2017 Jun 26;2(1):e10. doi: 10.2196/diabetes.6884. PMID 30291058
- See also: RENEWING HEALTH, REgioNs of Europe WorkINg toGether for HEALTH Click here for more information about this study:" — http://www.renewinghealth.eu/